CLINICAL TRIAL: NCT01982500
Title: A Multicentre, Observational Study of Bevacizumab (Avastin) Added to Front-line Chemotherapy in Patients With Stage IIIb, IIIC or IV Epithelial Ovarian Cancer, Fallopian Tube Carcinoma or Primary Peritoneal Carcinoma in Routine Clinical Practice.
Brief Title: Observation of Bevacizumab Plus Front-line Chemotherapy in Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CT/12.01
Record Dates: First submitted 2013-11-03; First posted 2013-11-13 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Chemotherapy; Anti-angiogenic agent; Bevacizumab; Front Line
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Avastin regimens: Patients who are going to receive chemotherapy plus Avastin (bevacizumab)

SUMMARY:
Investigators propose to assess,the safety and tolerability profile (number of participants with adverse events) of bevacizumab (Avastin) when added to chemotherapy as front-line treatment of epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma

DETAILED DESCRIPTION:
In the last decade, clinical studies with bevacizumab (Avastin) in various tumors have shown encouraging results in terms of efficacy/safety. However there is no data generated in Greek population with regards to safety and efficacy of bevacizumab in front line Ovarian Cancer. Two prior global phase III randomized trials showed that the addition of concurrent bevacizumab to standard chemotherapy and maintenance bevacizumab significantly increased the PFS in patients with advanced ovarian cancer It would be relevant to document the real life clinical data of bevacizumab in combination with chemotherapy (paclitaxel/carboplatin) in Front Line Ovarian Cancer as prescribed by the medical oncologists in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Histologically confirmed advanced stage III (suboptimally debulked >1cm of residual disease) or stage IV ovarian cancer fallopian tube carcinoma or primary peritoneal cancer following surgical debulking with the aim of maximal surgical cytoreduction
* One or more measurable lesions (≥1cm in diameter with spiral CT scan or ≥2cm with conventional techniques) according to RECIST criteria
* ECOG performance status ≤2
* Adequate haematological, renal and hepatic function
* Urine protein <2+ (dipstick)
* Life expectancy of >12 weeks

Exclusion Criteria:

* Previous front line treatment for ovarina cancer
* Previous radiotherapy to target lesions
* Patients with brain metastases and/or cancerous meningitis
* Presence or history of other neoplasm except properly treated basal cell skin cancer or in situ cervical carcinoma
* Patients participating in interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics for cancer prevention
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2016-10 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Every 3 weeks up to 18 weeks
  In this observational study investigators are going to assess standard schedules in which administration was every 3 weeks

SECONDARY OUTCOMES:
Number of Participants with Response Rate | Disease evaluation at Week 3
  In this observational study investigators are going to assess standard schedules in which the disease evaluation was performed every 3 weeks
Percentage of Patients with Progression Free Survival | 1 year
Patients Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Kalykaki, MD, Principal Investigator — Hellenic Oncology Research Group
Locations (6):
- Greece (6):
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dept. of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki